CLINICAL TRIAL: NCT00341250
Title: Randomized, Controlled, Phase 1/2 Study of the Safety and Immunogenicity of AMA1-C1/Alhydrogel Vaccine for Plasmodium Falciparum Malaria in Children in Doneguebougou and Bancoumana, Mali
Brief Title: Malaria Vaccine in Children in Mali
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: RCHSPB
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999906081; 06-I-N081
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-29

CONDITIONS: Malaria
Keywords: Blood Stage; Investigational; Endemic; Malaria
MeSH Terms: conditions — Malaria; Burkitt Lymphoma

INTERVENTIONS:
Drug: AMA1-C1/Alhydrogel Malaria Vaccine

SUMMARY:
This study will test an experimental vaccine called AMA1-C1 in children to see if it is safe and if it reduces episodes of malaria parasitemia (parasites in the blood) in children exposed to malaria. Malaria affects about 300 million to 500 million people worldwide each year, causing from 2 million to 3 million deaths, mostly among children less than 5 in sub-Saharan Africa. It is the leading cause of death and illness among the general population of Mali in West Africa. Increasing drug resistance to the malaria parasite and widespread resistance of mosquitoes (the insects that transmit the parasite) to pesticides are reducing the ability to control malaria through these strategies. A vaccine that could reduce illness and death from malaria would be a valuable new resource in the fight against this disease. AMA1-C1 is an experimental vaccine developed by the NIAID. Tests of AMA1-C1 in 87 healthy people in the United States and in Mali found no serious harmful side effects of the vaccine.

Two- and three-year-old children who live in Don gu bougou or Bancoumana, Mali, and are in general good health may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood and urine tests.

Participants are randomly assigned to receive two injections (shots) of either AMA1-C1 or a Haemophilus influenzae type B vaccine called Hiberix® (Registered Trademark), which is approved and used in Mali. All shots are given in the thigh muscle. Before the first shot, a small blood sample is obtained to make sure the child is well and to see if he or she has antibodies to the malaria parasite. The second shot is given 4 weeks after the first. After each shot, participants are observed in the clinic for 30 minutes. They return to the clinic 1, 2, 3, 7 and 14 days after each shot for a physical examination. Blood samples are drawn at some visits to check for side effects of the vaccine and to measure the response to it.

During the rainy season after the second vaccination, subjects come to the clinic once a month for an examination. Any child who has been ill with a disease that could be malaria has a blood sample collected by fingerstick to test for malaria and to learn about the malaria parasites causing the infection. Every fourth visit a fingerstick sample is taken regardless of whether the child has been sick. If a child becomes sick at any time during the study, he or she will be brought to the clinic for examination a...

DETAILED DESCRIPTION:
Apical membrane antigen-1 (AMA1) is a surface protein expressed during the asexual blood stage of P. falciparum. It is produced as an 83-kDa polypeptide by mature schizonts in infected erythrocytes. In clinical studies in malaria-unexposed adults in the USA and in malaria-exposed adults in Mali, AMA1-C1/Alhydrogel was safe and immunogenic. This study will evaluate its safety and immunogenicity in malaria-exposed children living in an area of seasonal malaria transmission.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males or females aged 2 to less than 4 years old. Children must be born no earlier than September 1, 2002 and must have had their second birthday prior to first vaccination.

Known residents of the village of Doneguebougou, Mali or Bancoumana.

Good general health as determined by means of the screening procedures.

Available for the duration of the trial (52 weeks).

Willingness to participate in the study as evidenced by parents/legal guardians signing or fingerprinting the informed consent document.

EXCLUSION CRITERIA:

Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, chronic infectious or renal disease by history, physical examination, and/or laboratory studies including urinalysis.

Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer or the parent/legal guardian to understand and cooperate with the study protocol.

Laboratory evidence of liver disease (alanine aminotransferase (ALT) greater than 1.25 times the upper limit of normal of the testing laboratory).

Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory, or more than trace protein or blood on urine dipstick testing).

Laboratory evidence of hematologic disease (absolute leukocyte count less than 3000/mm(3) or greater than 14,500/mm(3), absolute lymphocyte count less than 1000/mm(3), platelet count less 120,000/mm(3), or hemoglobin less than 8.5 g/dL).

Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

Participation in another investigational vaccine or drug trial within 30 days of starting this study, or while this study is ongoing.

History of a severe allergic reaction or anaphylaxis.

Severe asthma (emergency room visit or hospitalization within the last 6 months).

Positive ELISA for HCV.

Positive HBsAg by ELISA.

Known immunodeficiency syndrome.

Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study.

Receipt of a live vaccine within past 4 weeks (e.g. measles/mumps/rubella (MMR)) or a non-live vaccine (e.g. diphtheria/pertussis/tetanus (DPT)) within past 2 weeks prior to entry into the study.

History of a surgical splenectomy.

Receipt of a blood transfusion within the past 6 months.

Previous receipt of an investigational malaria vaccine.

History of a known allergy to nickel.

History of known allergy to yeast.

Known hypersensitivity to any component of the Hib vaccine (tetanus toxoid, lactose).

Previous administration of Hib vaccines.

Known thrombocytopenia or bleeding disorders.

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900
Dates: Start 2006-01-19; Study Completion 2006-12-08

CONTACTS AND LOCATIONS:
Locations (2):
- Mali (2):
  - Bancoumana Clinical Trial Center, Bankoumana
  - Doneguebougou Malaria Vaccine Center, Donéguébougou

REFERENCES:
- [Background] Narum DL, Thomas AW. Differential localization of full-length and processed forms of PF83/AMA-1 an apical membrane antigen of Plasmodium falciparum merozoites. Mol Biochem Parasitol. 1994 Sep;67(1):59-68. doi: 10.1016/0166-6851(94)90096-5. PMID 7838184
- [Background] Crewther PE, Culvenor JG, Silva A, Cooper JA, Anders RF. Plasmodium falciparum: two antigens of similar size are located in different compartments of the rhoptry. Exp Parasitol. 1990 Feb;70(2):193-206. doi: 10.1016/0014-4894(90)90100-q. PMID 2404781
- [Background] Waters AP, Thomas AW, Deans JA, Mitchell GH, Hudson DE, Miller LH, McCutchan TF, Cohen S. A merozoite receptor protein from Plasmodium knowlesi is highly conserved and distributed throughout Plasmodium. J Biol Chem. 1990 Oct 15;265(29):17974-9. PMID 2211675
- [Derived] Dicko A, Sagara I, Ellis RD, Miura K, Guindo O, Kamate B, Sogoba M, Niambele MB, Sissoko M, Baby M, Dolo A, Mullen GE, Fay MP, Pierce M, Diallo DA, Saul A, Miller LH, Doumbo OK. Phase 1 study of a combination AMA1 blood stage malaria vaccine in Malian children. PLoS One. 2008 Feb 13;3(2):e1563. doi: 10.1371/journal.pone.0001563. PMID 18270560